CLINICAL TRIAL: NCT06258291
Title: A Multi-center Randomized Controlled First in Human Trial to Assess the Feasibility and Preliminary Safety Data of Adjunctive Treatment with the HemoSystem REBOOT in Critically Ill PatientS with Sepsis-induced ImmunOsuppREssion (RESTORE I)
Brief Title: First in Human Trial to Assess the Feasibility and Preliminary Safety of Adjunctive Treatment with the HemoSystem REBOOT in Critically Ill Patients with Sepsis-induced Immunosuppression
Acronym: RESTORE I
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: hemotune AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Restore I; HNT001 (Other: hemotune AG)
Record Dates: First submitted 2024-01-12; First posted 2024-02-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Septic Shock
Keywords: immunosuppression
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: randomized controlled trial: treatment in addition to standard of care versus standard of care alone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Experimental): The REBOOT Hemosystem will be tested in the treatment arm for a maximum of 5 treatments, the treatment will be applied in addition to standard of care alone.
  Interventions: Device: Hemosystem REBOOT
- Standard of care (No Intervention): Best standard of care will be applied to these patients.

INTERVENTIONS:
Device: Hemosystem REBOOT — The HemoSystem REBOOT will selectively remove three mediators largely contributing to sepsis-induced immunosuppression, from extracorporeal circulation based on magnetic beads.
  Other Names: extracorporeal blood purification
  Arms: Treatment arm

SUMMARY:
The aim of this randomized controlled trial is to restore immune function by selectively removing three mediators largely contributing to sepsis-induced immunosuppression from extracorporeal circulation.

DETAILED DESCRIPTION:
The treatment safety and the kinetics of specific biomarkers will be assessed to evaluate the selection of the treatment regimen. In a first step, 16 patients will be randomized 1:1 into two arms:

Treatment arm 1: One treatment of 2 hours per day for a maximum of five days or until ICU discharge or death or withdrawal of consent, whichever occurs first.

Control arm: Five consecutive days following the first mHLA-DR measurement post study randomization, or until ICU discharge or death or withdrawal of consent, whichever occurs first

And the end of this treatment phase, it will be decided whether the dosage regimen of HemoSystem REBOOT needs to be adapted and another eight patients have to be enrolled with 2 treatments per day, and a maximum of five treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Written informed consent according to national requirements.
3. Hospitalized in ICU or IMC at randomization.
4. Expected length of intensive care unit stay (from randomization) >48 hours.
5. Suspected or confirmed bacterial sepsis.
6. Septic shock diagnosis at any time during ICU/IMC stay according to Sepsis - 3 criteria definition:

   1. an infection (suspected or confirmed);
   2. persisting hypotension requiring any dose of vasopressors (norepinephrine, vasopressin) to maintain a systemic mean blood pressure > 65 mmHg despite adequate fluid resuscitation (minimum of 30 ml/kg crystalloids);
   3. elevated lactate ≥ 2.0 mmol/L with suspected hypoperfusion.
7. Persistent immunosuppression defined as mHLA-DR expression levels < 5600 Ab/cell (Cyto-Chex tubes) in at least two consecutive measurements 20-72 hours apart.

Exclusion criteria:

1. Current ongoing chronic treatment using immunosuppressive biologicals or active lymphocyte therapy (e.g. endoxan, rituximab) or corticosteroid use at a dose > 10 mg/day equivalent of prednisone. However, acute treatment using a maximum dose of hydrocortisone of 200 mg/day for sepsis is allowed.
2. Patient with preexisting known severe immune deficiency (e.g. severe combined immunodeficiency, HIV infection, AIDS).
3. Active or planned extracorporeal membrane oxygenation treatment.
4. Active or planned other extracorporeal blood purification treatments with systems like CytoSorb®, ToraymyxinTM, Gambro Adsorba, etc.
5. Patients post solid-organ transplantation.
6. Known active malignancy (i.e. patients under active anti-malignant treatment).
7. Acute severe burn injury > 20% of the body surface area.
8. Contraindication to use the HemoSystem:

   1. Sensitivity / allergy to HemoSystem components
   2. Body weight < 50 kg
   3. Platelets count < 20,000/µL
   4. History of heparin-induced thrombocytopenia.
9. Females who are known to be pregnant or known to be breastfeeding (b-HCG testing performed in female patients aged < 55 years),
10. Moribund patient with life expectancy < 48h
11. Known history of bleeding disorders or severe coagulopathies (e.g., Hemophilia A, Hemophilia B, Idiopathic Thrombocytopenic Purpura, Von Willebrand Disease types I, II, and III)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-28 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Biomarker for sepsis induced immunosuppression (monocytic HLA-DR = mHLA-DR) | pre-procedure immune marker levels compared to post-treatment levels at least 24 hours after last treatment (on average estimated day 6 after treatment start)
  Change in mHLA-DR levels during treatment compared to the standard of care arm alone

SECONDARY OUTCOMES:
To determine all-cause mortality up to 90 days follow-up | through the end of the study (on average 90 days follow up)
  Difference in mortality between treatment arm and standard of care arm
Need for organ support therapy (the number of days on organ support in the intensive care unit (index admission) defined by (1) invasive mechanical ventilation, (2) Intermittent or continuous renal replacement therapy, (3) any vasopressor support. | until the end of the initial ICU admission (on average day 10 after initial ICU admission)
  Difference between treatment arm and standard of care arm
To assess the total number of organ support free days in intensive and intermediate care unit | until the end of the initial ICU admission (on average day 10 after initial ICU admission)
  Difference in total number of organ support free days between treatment arm and standard of care arm
To assess the change of Sequential Organ Failure Assessment (SOFA) score (ranging from 0 =normal to 4=significantly impaired per category) | through the end of the study (on average 90 days follow up)
  Difference in SOFA score between treatment arm and standard of care arm
To assess vasopressor doses during intensive and intermediate care unit stay | until the end of the initial ICU admission (on average day 10 after initial ICU admission)
  To assess the difference in dosing between the treatment arm and standard of care arm
To assess the use of antimicrobial medication | through the end of the study (on average 90 days follow up)
  Difference in days on antimicrobials vs days off antimicrobials between treatment arm and standard of care arm
To evaluate the change in the biomarker (for sepsis-induced immunosuppression) mHLA-DR concentration at various timepoints during ICU stay | at admission to ICU, on the day of first, 2nd, 3rd, 4th, and 5th treatment, and daily up to 72 hours after last treatment.
  Difference in immune markers between treatment arm and standard of care arm will be compared
To assess the technical success of in vivo target removal | immediately after last treatment
  Technical success rate in treatment arm
Number of SADEs in treatment arm | through the end of the study (on average 90 days follow up)
  SADE rate

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Schefold, Prof, Principal Investigator — University Hospital Berne, Inselspital
Locations (2):
- Switzerland (2):
  - University Hospital Bern Inselspital, Bern
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No